CLINICAL TRIAL: NCT03272529
Title: Comparative Effectiveness of Patient-Specific Simulated Rehearsal for Percutaneous Nephrolithotomy (PCNL)
Brief Title: Simulated Rehearsal for Percutaneous Nephrolithotomy
Acronym: PCNL
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ahmed Ghazi, Assistant Professor, University of Rochester
Other Study IDs: 68871
Record Dates: First submitted 2017-08-22; First posted 2017-09-05 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Nephrolithotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient-specific simulated rehearsals: Participants recruited to this cohort will complete just-in-time simulation, i.e., practice a short time prior to the live event using hydrogel models designed from patients' imaging, incorporating the necessary anatomy, physiology, and pathology specific to each patient. This is in addition to standard prerequisite simulation training.
  Interventions: Other: Patient-specific simulated rehearsals
- Idealized simulated rehearsals: Participants recruited to this cohort will complete just-in-time simulation, i.e., practice a short time prior to the live event using hydrogel models that incorporate the necessary anatomy, physiology, and pathology of an ideal training case. This is in addition to standard prerequisite simulation training.
  Interventions: Other: Idealized simulated rehearsals
- Standard simulation: Participants recruited to this cohort will only have completed the standard prerequisite simulation training similar to the two other groups (didactic lecture, hands-on simulation training to proficiency and live case observation), that represents the current standard of care. No further simulation would be conducted in this group in addition to the standard.
  Interventions: Other: Standard simulation

INTERVENTIONS:
Other: Patient-specific simulated rehearsals — Using 3-D printing and polymer technology, the investigators' team will construct patient-specific simulated hydrogel models designed from patients' imaging, incorporating the necessary anatomy, physiology, and pathology specific to each patient. These models will be constructed at the Simulation Innovation laboratory within the Department of Urology, University of Rochester. The process involves importing DICOM files of patient participants C.T. scans into 3D processing software, creating virtual models of kidney parenchyma incorporating the kidney, urinary system, stone and abdominal wall. Surgical phantoms are then created using 3D printing and polymer hydrogels, to recreate the entire procedure.
  Groups: Patient-specific simulated rehearsals
Other: Idealized simulated rehearsals — Using 3D printing and polymer technology, the investigators' team will construct a validated generic simulated hydrogel model with a complex kidney stone, incorporating the necessary anatomy, physiology and pathology. These models will be constructed at the Simulation Innovation laboratory within the department of urology at the University of Rochester. Generic models incorporating the kidney, PCS, staghorn stone, abdominal wall, and other relevant anatomical elements (bowel, perinephric fat, solid organs and bony structures) will be constructed. Participants in his group will complete the simulation replicating all steps of the procedure of this ideal training case that is not specific to a particular patient.
  Groups: Idealized simulated rehearsals
Other: Standard simulation — Participants recruited to this cohort will only have completed the standard prerequisite simulation training similar to the two other groups (didactic lecture, hands-on simulation training to proficiency and live case observation), that represents the current standard of care. No further simulation would be conducted in participants of this group in addition to the standard.
  Groups: Standard simulation

SUMMARY:
Surgical simulation provides opportunities for surgeons to practice specific skills, prior to performing complex tasks on patients, with the goal of reducing potential errors and providing a safer procedure for the patient. The investigators will use a novel approach to simulation (patient-specific rehearsals) i.e., practice a short time prior to the live event that uses gel models of organs created by a 3D printer, and that are specific to each patient versus models that represent an ideal training model. The investigators' overarching goals are to improve patient outcomes by developing the best platform for surgeons to efficiently enhance performance prior to live surgery.

DETAILED DESCRIPTION:
Surgical simulation provides opportunities for both medical residents and expert surgeons to practice specific skills, prior to performing complex tasks on patients, with the goal of reducing potential errors and providing a safer procedure for the patient. Most studies have addressed surgical simulation carried out in dry and animation laboratories at a significantly different time than the actual surgery on patients. For most surgeons-in-training, there is no intermediate stage between practice and performance. Learning takes place in isolation, and surgeons do not routinely experience how dexterity skills are affected by context until they perform an actual operation. The investigators will use a unique approach to simulation (just-in-time simulation i.e., practicing in close proximity to live surgery). The investigators believe that this approach will be most beneficial for highly technical procedures such as Percutaneous Nephrolithotomy (PCNL), because this approach could familiarize the surgeon with the case, enable them to try different approaches, identify potential dangers, and even optimize the selection of tools for the procedure. This type of simulation is usually performed using idealized or generic models that can improve a surgeon's technical, cognitive, and hand - eye coordination performance, of this specific procedure prior to the live surgery but is not personalized for an individual patient.

The investigators' efforts at the Simulation Innovation Laboratory (SIL) at the University of Rochester in combining 3D printing technology with polymer research has provided a platform for reproducing patient specific water-based gel models with accurate portrayal of anatomical characteristics including individual patient variations, but also with the capacity to reproduce tissue characteristics and replicate the comprehensive operative experience. Patient specific simulations, however, allow surgeons to practice, plan and address potential problems related to a specific patient's surgery before performing the actual surgery. The investigators developed three-dimensional (3D) models, which reproduce patient-specific anatomy and tissue characteristics, allowing for a rehearsal that is an accurate representation of an actual procedure to be done, in this case Percutaneous Nephrolithotomy for the treatment of complex renal stones.

In the present era of simulation, no standard form of simulation exists that is performed directly prior to the live surgery, nor is there any form of personalized simulation for each patient. In this study the investigators aim to compare just-in-time simulation using either patient-specific or idealized training models and compare their impact on operative performance following Percutaneous Nephrolithotomy (PCNL). Secondary objectives are to assess their impact on patient outcomes following PCNL. The investigators overarching goals are to improve patient outcomes by developing the best platform for surgeons to efficiently enhance their performance prior to live surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to undergo PCNL surgery at the University of Rochester Medical Center
* Ability to give informed consent
* Willing to participate in the study
* Any racial or ethnic origin

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is comprised of 100 PCNL patients, 2 faculty expert urologists, and 12 urology trainees selected from years PGY3 and above.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Fluoroscopy time measured during percutaneous nephrolithotomy (PCNL) | At the end of each surgical procedure, approximately 24 hours after surgery
  Fluoroscopy time is reported on completion of PCNL, the metric will be measured in minutes as a continuous variable.
Percutaneous access (PCA) attempts | At the end of each surgical procedure, approximately 24 hours after surgery
  PCA attempts is reported on completion of the PCNL, the metric will be measured in number of attempts as a continuous variable.
Surgical complications | From date of surgery up to 30 days postoperative, every complication encountered during that time will be recorded
  Intraoperative and postoperative complications will be measured and reported using the modified Clavien-Dindo classification of surgical complications (Grade 1 to 5).
Objective evaluation of surgical performance (Virtual percutaneous nephrostolithotomy GRS) | At the end of each surgical procedure, approximately 24 hours after surgery
  All surgical cases will be recorded and reviewed by expert surgeons using a tool that specializes in evaluation of PCNL surgical performance, the Virtual percutaneous nephrostolithotomy GRS (a validated assessment of percutaneous Nephrolithotomy using a 5-point Likert-type scale, of 5 domains including knowledge of renal anatomy, trajectory planning, instrument use, need for instructor assistance and overall task performance), these will be measured as a continuous variable.
Surgeon take-over | At the end of each surgical procedure, approximately 24 hours after surgery
  Surgeon take-over is reported on completion of the PCNL; the metric will be measured as a nominal variable (yes or no) when the surgeon in the operating room takes over the case.
Change in the volume of stone before and after PCNL surgery (Stone clearance) | Zero at date of randomization and serial measurements at 1 and up to 30 days after surgery
  The difference between preoperative (within a month prior to surgery) and postoperative (1-30 days after surgery) in millimeters using imaging techniques (KUB, Ultrasound and CT-IVP).

SECONDARY OUTCOMES:
Change in the volume of ratio of red blood cells to total blood volume (HCT) | Zero at date of randomization and serial measurements at 12 and 24 hours after surgery
  The difference between preoperative (within a week prior to surgery) and postoperative (12 and 24 hours after surgery) using the blood test HCT.
Hospital stay | From date of admission up to 30 days after surgery
  The length of hospital stay will be measured from time of admission to day of discharge and will be reported in days
Hospital readmission | From date of surgery up to 30 days postoperative, every hospital readmission encountered during that time will be recorded
  The readmission rates of patients enrolled in the study will be measured and reported in number of patients
Blood transfusion | From date of randomization up to 30 days after surgery every unit of blood transfused during that time will be recorded
  The presence or absence (+/-) and how many units will be measured (blood units)
Change in postoperative renal functions | Zero at date of randomization and serial measurements at 12 hours , 1 day and 30 days after surgery
  The difference between preoperative (within a week prior to surgery) and postoperative (12 hours, 1 day and 30 days after surgery) using estimated GFR measured through serum creatinine blood test.
Additional stone procedures | From date of surgery up to 30 days postoperative, every additional procedure performed during that time will be recorded
  The presence or absence (+/-) and how many additonal procedures to achieve complete stone clearance after the procedure will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ghazi, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No